CLINICAL TRIAL: NCT02828839
Title: Prostate Biopsy Access Needle & Needle Guide Feasibility Study
Acronym: STABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perineologic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P-101
Record Dates: First submitted 2016-06-30; First posted 2016-07-12 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: Transperineal; Transrectal; Needle Guide; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive standard of care prostate biopsies through the use of a trans-rectal ultrasound probe for needle placement and guidance. The intervention for all patients receiving a prostate biopsy will include the use of an investigational single use, disposable stainless steel access needle and a single use, disposable polymeric needle guide.
  Interventions: Procedure: Access needle

INTERVENTIONS:
Procedure: Access needle — The primary purpose of the single-use disposable access needle is to guide the use of a biopsy gun to obtain a tissue sample from the patient's prostate gland through a percutaneous puncture of the perineum. The primary purpose of the disposable needle guide is to stabilize the needle biopsy and better approximate the most direct path to the prostate.

SUMMARY:
The objective of the study is to assess the design features of a modified stainless steel access needle (single use disposable) in a clinical setting and a disposable, single use, custom-made, polymer needle guide used in conjunction with a rectal ultrasound probe. The disposable stainless steel access needle may be used with or without the disposable needle guide, but will always be used with ultrasound image guidance and a biopsy gun. The primary purpose of the single-use disposable access needle is to guide the use of a biopsy gun to obtain a tissue sample from the patient's prostate gland through a percutaneous puncture of the perineum. The primary purpose of the disposable needle guide is to stabilize the needle biopsy and better approximate the most direct path to the prostate.

DETAILED DESCRIPTION:
The objective of the study is to assess the design features of a modified stainless steel access needle (single use disposable) in a clinical setting with and a disposable, single use, custom-made, polymer needle guide used in conjunction with a rectal ultrasound probe. The disposable stainless steel access needle may be used with or without the disposable needle guide, but will always be used with ultrasound image guidance and a biopsy gun. The primary purpose of the single-use disposable access needle is to guide the use of a biopsy gun to obtain a tissue sample from the patient's prostate gland through a percutaneous puncture of the perineum. The primary purpose of the disposable needle guide is to stabilize the needle biopsy and better approximate the most direct path to the prostate. For some subjects, the study will assess the fit and functionality of the stainless steel access needle when used in conjunction with the disposable needle guide as well as multiple handling aspects of the access needle and disposable needle guide when utilized in a prostate biopsy procedure. The study will also assess the ability of trans-rectal ultrasound to appropriately image the stainless steel access needle and biopsy gun needle at, near, and within the prostate tissue.

ELIGIBILITY:
Inclusion Criteria:

* Males requiring a needle-biopsy of the prostate with ultrasound assistance via a trans-rectal ultrasound probe
* Otherwise healthy patient with no serious acute or chronic illness

Exclusion Criteria:

* Patients with a partial or complete prostectomy
* Patients with active infection of the prostate, perineum, rectum, bowel, or peritoneum
* Patients with serious acute or chronic illness
* Cannot read and comprehend simple instructions in English
* Poorly controlled psychiatric disease
* Females

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the handling characteristics of the access needle and needle guide. | The time point at which this will be measured is at the end of the prostate biopsy procedure up to 30 days through study completion.
  Assessment of the handling characteristics of the single use, disposable stainless steel access needle and the single use, disposable polymeric needle guide will be completed by the user completing a questionnaire rating various performance characteristics of the access needle and the needle guide at the completion of each prostate biopsy. Using a scale from 1 to 5, with 1 being poor and 5 being excellent, each characteristic of the access needle and the needle will be rated. The results will be summarized across all characteristics and reported as percentages of each rating scale indicator, 1 through 5.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Allaway, DO, Study Director — Perineologic
Locations (1):
- Corbin Clinical Resources, Cumberland, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rodriguez LV, Terris MK. Risks and complications of transrectal ultrasound guided prostate needle biopsy: a prospective study and review of the literature. J Urol. 1998 Dec;160(6 Pt 1):2115-20. doi: 10.1097/00005392-199812010-00045. PMID 9817335
- [Background] Emiliozzi P, Corsetti A, Tassi B, Federico G, Martini M, Pansadoro V. Best approach for prostate cancer detection: a prospective study on transperineal versus transrectal six-core prostate biopsy. Urology. 2003 May;61(5):961-6. doi: 10.1016/s0090-4295(02)02551-7. PMID 12736016
- See also: Perineologic approach to prostate biopsies — http://www.perineologic.com